CLINICAL TRIAL: NCT01562275
Title: A Phase Ib, Open-Label, Dose-Escalation Study of the Safety, Tolerability and Pharmacokinetics of GDC-0973 and GDC-0068 in Patients With Locally Advanced or Metastatic Solid Tumors
Brief Title: A Study Evaluating the Safety, Tolerability, and Pharmacokinetics of GDC-0973 in Combination With GDC-0068 When Administered in Participants With Locally Advanced or Metastatic Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GE28079; 2012-003934-18 (EudraCT Number)
Record Dates: First submitted 2012-03-21; First posted 2012-03-23 (Estimated); Results first posted 2016-03-28 (Estimated); Last update posted 2016-03-28 (Estimated); Status verified 2016-02

CONDITIONS: Neoplasms
Keywords: GDC0973; MEK; MEK inhibitor; GDC0068; Akt; Akt inhibitor
MeSH Terms: conditions — Neoplasms | interventions — ipatasertib; cobimetinib

ARMS (3):
- Dose escalation stage 1 (Arm A): Cobimetinib and Ipatasertib (Experimental): Participants will receive cobimetinib (GDC-0973) capsules (at a starting dose of 40 mg) and ipatasertib (GDC-0068) capsules (at a starting dose of 200 mg) from Days 1 to 21 and then 7 days off study drugs from Days 22 to 28 in continuous 28-day cycles. Doses will be increased to identify maximum tolerated dose (MTD) or potential recommended Phase 2 dose (RP2D). Treatment will continue until disease progression, unacceptable toxicity, or any other discontinuation criterion meets.
  Interventions: Drug: Ipatasertib; Drug: Cobimetinib
- Dose escalation stage 1 (Arm B): Cobimetinib and Ipatasertib (Experimental): Participants will receive cobimetinib (GDC-0973) capsules (at a starting dose of 100 mg) on Days 1, 4, 8, 11, 15, and 18 and ipatasertib (GDC-0068) capsules (at a starting dose of 200 mg) from Days 1 to 21 and then 7 days off study drugs from Days 22 to 28 in continuous 28-day cycles. Doses will be increased to identify MTD or potential RP2D. Treatment will continue until disease progression, unacceptable toxicity, or any other discontinuation criterion meets.
  Interventions: Drug: Ipatasertib; Drug: Cobimetinib
- Stage 2 (Indication specific dose expansion cohort) (Experimental): Participants will receive cobimetinib (GDC-0973) capsules on Days 1, 4, 8, 11, 15, and 18 and ipatasertib (GDC-0068) capsules from Days 1 to 21 and then 7 days off study drugs from Days 22 to 28 in continuous 28-day cycles, at doses identified as MTD/potential RP2D from Stage 1. Treatment will continue until disease progression, unacceptable toxicity, or any other discontinuation criterion meets. This indication specific cohort will include participants with phosphatase and tensin homolog (PTEN)-loss triple-negative breast cancer and PTEN-loss endometrial carcinoma.
  Interventions: Drug: Ipatasertib; Drug: Cobimetinib

INTERVENTIONS:
Drug: Ipatasertib — multiple doses
  Other Names: GDC-0068
Drug: Cobimetinib — multiple doses
  Other Names: GDC-0973

SUMMARY:
This open-label, multicenter, Phase Ib dose-escalation study will evaluate the safety, tolerability and pharmacokinetics of oral dosing of GDC-0973 and GDC-0068 administered in combination in patients with locally advanced or metastatic solid tumors. Cohorts of patients will receive multiple ascending doses of GDC-0973 and GDC-0068. Anticipated time on study treatment is until disease progression or unacceptable toxicity occurs.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically documented locally advanced or metastatic solid tumors for which standard therapies either do not exist or have proven ineffective or intolerable
* Evaluable disease or disease measurable per Response Evaluation Criteria in Solid Tumors (RECIST)
* Life expectancy >/= 12 weeks
* Adequate hematologic and end organ function

Exclusion Criteria:

* History of prior significant toxicity from another MEK pathway inhibitor requiring discontinuation of treatment
* History of prior significant toxicity from another phosphoinositide 3-kinase (PI3K) or Akt pathway or mammalian target of rapamycin (mTOR) inhibitor requiring discontinuation of treatment
* Anti-cancer therapy within 28 days prior to first dose of study drug, except as stated in protocol
* History of type I or type II diabetes mellitus requiring insulin
* Current severe, uncontrolled systemic disease (e.g. clinically significant cardiovascular, pulmonary, or metabolic disease)
* Clinically significant history of liver disease, current alcohol abuse, or current known active infection with HIV, hepatitis B or hepatitis C virus
* Active autoimmune disease
* Pregnant or lactating women
* Known brain metastases that are untreated, symptomatic, or require therapy to control symptoms
* History of glaucoma
* History of retinal vein occlusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2012-04; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Genentech, Inc.
Locations (5):
- United States (3):
  - Boston, Massachusetts
  - Detroit, Michigan
  - Nashville, Tennessee
- Spain (2):
  - Barcelona, Barcelona
  - Valencia, Valencia

REFERENCES:
- [Derived] Shapiro GI, LoRusso P, Cho DC, Musib L, Yan Y, Wongchenko M, Chang I, Patel P, Chan IT, Sanabria-Bohorquez S, Meng RD, Bendell JC. A phase Ib open-label dose escalation study of the safety, pharmacokinetics, and pharmacodynamics of cobimetinib (GDC-0973) and ipatasertib (GDC-0068) in patients with locally advanced or metastatic solid tumors. Invest New Drugs. 2021 Feb;39(1):163-174. doi: 10.1007/s10637-020-00975-6. Epub 2020 Jul 31. PMID 32737717

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Study included two stages. Stage 1: dose escalation cohorts (DEC), consisted of Arm A (concurrent 21 day dosing followed by 7 day dosing holiday) and Arm B (intermittent dosing). Stage 2: indication specific expansion cohorts (PTEN-low endometrial carcinoma and PTEN-low triple-negative breast cancer) treated with recommended phase 2 dose.
Groups:
- DEC Arm A: 40 mg Cobimetinib + 200 mg Ipatasertib: Participants received oral 40 milligrams (mg) cobimetinib and 200 mg ipatasertib concurrently once daily on Days 1-21, with a 7-day dosing holiday on Days 22-28, every 28 days (1 Cycle=28 Days) until disease progression, unacceptable toxicity, or any other discontinuation criteria were met.
- DEC Arm A: 60 mg Cobimetinib + 200 mg Ipatasertib: Participants received oral 60 mg cobimetinib and 200 mg ipatasertib concurrently once daily on Days 1-21, with a 7-day dosing holiday on Days 22-28, every 28 days (1 Cycle=28 Days) until disease progression, unacceptable toxicity, or any other discontinuation criteria were met.
- DEC Arm A: 60 mg Cobimetinib + 300 mg Ipatasertib: Participants received oral 60 mg cobimetinib and 300 mg ipatasertib concurrently once daily on Days 1-21, with a 7-day dosing holiday on Days 22-28, every 28 days (1 Cycle=28 Days) until disease progression, unacceptable toxicity, or any other discontinuation criteria were met.
- DEC Arm A: 40 mg Cobimetinib + 400 mg Ipatasertib: Participants received oral 40 mg cobimetinib and 400 mg ipatasertib concurrently once daily on Days 1-21, with a 7-day dosing holiday on Days 22-28, every 28 days (1 Cycle=28 Days) until disease progression, unacceptable toxicity, or any other discontinuation criteria were met.
- DEC Arm B: 100 mg Cobimetinib + 200 mg Ipatasertib: Participants received oral 200 mg ipatasertib once daily on Days 1-21 consecutively with concurrent dosing of 100 mg cobimetinib on Days 1, 4, 8, 11, 15, and 18 with a 7-day dosing holiday on Days 22-28, every 28 days (1 Cycle=28 Days) until disease progression, unacceptable toxicity, or any other discontinuation criteria were met.
- DEC Arm B: 125 mg Cobimetinib + 200 mg Ipatasertib: Participants received oral 200 mg ipatasertib once daily on Days 1-21 consecutively with concurrent dosing of 125 mg cobimetinib on Days 1, 4, 8, 11, 15, and 18 with a 7-day dosing holiday on Days 22-28, every 28 days (1 Cycle=28 Days) until disease progression, unacceptable toxicity, or any other discontinuation criteria were met.
- DEC Arm B: 125 mg Cobimetinib + 400 mg Ipatasertib: Participants received oral 400 mg ipatasertib once daily on Days 1-21 consecutively with concurrent dosing of 125 mg cobimetinib on Days 1, 4, 8, 11, 15, and 18 with a 7-day dosing holiday on Days 22-28, every 28 days (1 Cycle=28 Days) until disease progression, unacceptable toxicity, or any other discontinuation criteria were met.
- DEC Arm B: 150 mg Cobimetinib + 300 mg Ipatasertib: Participants received oral 300 mg ipatasertib once daily on Days 1-21 consecutively with concurrent dosing of 150 mg cobimetinib on Days 1, 4, 8, 11, 15, and 18 with a 7-day dosing holiday on Days 22-28, every 28 days (1 Cycle=28 Days) until disease progression, unacceptable toxicity, or any other discontinuation criteria were met.
- DEC Arm B: 175 mg Cobimetinib + 200 mg Ipatasertib: Participants received oral 200 mg ipatasertib once daily on Days 1-21 consecutively with concurrent dosing of 175 mg cobimetinib on Days 1, 4, 8, 11, 15, and 18 with a 7-day dosing holiday on Days 22-28, every 28 days (1 Cycle=28 Days) until disease progression, unacceptable toxicity, or any other discontinuation criteria were met.
- DEC Arm B: 150 mg Cobimetinib + 200 mg Ipatasertib: Participants received oral 200 mg ipatasertib once daily on Days 1-21 consecutively with concurrent dosing of 150 mg cobimetinib on Days 1, 4, 8, 11, 15, and 18 with a 7-day dosing holiday on Days 22-28, every 28 days (1 Cycle=28 Days) until disease progression, unacceptable toxicity, or any other discontinuation criteria were met.
- DEC Arm B: 100 mg Cobimetinib + 400 mg Ipatasertib: Participants received oral 400 mg ipatasertib once daily on Days 1-21 consecutively with concurrent dosing of 100 mg cobimetinib on Days 1, 4, 8, 11, 15, and 18 with a 7-day dosing holiday on Days 22-28, every 28 days (1 Cycle=28 Days) until disease progression, unacceptable toxicity, or any other discontinuation criteria were met.
- Endometrial Carcinoma: 140 mg Cobimetinib + 300 mg Ipatasertib: Participants with endometrial carcinoma received oral 300 mg ipatasertib once daily on Days 1-21 consecutively with concurrent dosing of 140 mg cobimetinib on Days 1, 4, 8, 11, 15, and 18 with a 7-day dosing holiday on Days 22-28, every 28 days (1 Cycle=28 Days) until disease progression, unacceptable toxicity, or any other discontinuation criteria were met.
- Breast Cancer: 140 mg Cobimetinib + 300 mg Ipatasertib: Participants with triple negative breast cancer received oral 300 mg ipatasertib once daily on Days 1-21 consecutively with concurrent dosing of 140 mg cobimetinib on Days 1, 4, 8, 11, 15, and 18 with a 7-day dosing holiday on Days 22-28, every 28 days (1 Cycle=28 Days) until disease progression, unacceptable toxicity, or any other discontinuation criteria were met.
Period: Stage 1
Arm/Group | DEC Arm A: 40 mg Cobimetinib + 200 mg Ipatasertib | DEC Arm A: 60 mg Cobimetinib + 200 mg Ipatasertib | DEC Arm A: 60 mg Cobimetinib + 300 mg Ipatasertib | DEC Arm A: 40 mg Cobimetinib + 400 mg Ipatasertib | DEC Arm B: 100 mg Cobimetinib + 200 mg Ipatasertib | DEC Arm B: 125 mg Cobimetinib + 200 mg Ipatasertib | DEC Arm B: 125 mg Cobimetinib + 400 mg Ipatasertib | DEC Arm B: 150 mg Cobimetinib + 300 mg Ipatasertib | DEC Arm B: 175 mg Cobimetinib + 200 mg Ipatasertib | DEC Arm B: 150 mg Cobimetinib + 200 mg Ipatasertib | DEC Arm B: 100 mg Cobimetinib + 400 mg Ipatasertib | Endometrial Carcinoma: 140 mg Cobimetinib + 300 mg Ipatasertib | Breast Cancer: 140 mg Cobimetinib + 300 mg Ipatasertib
Started | 3 | 7 | 3 | 4 | 4 | 4 | 3 | 7 | 3 | 7 | 3 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 7 | 3 | 4 | 4 | 4 | 3 | 7 | 3 | 7 | 3 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Death | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Non Compliance | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Progression of Disease | 2 | 6 | 2 | 1 | 2 | 4 | 1 | 7 | 2 | 5 | 3 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Period: Stage 2
Arm/Group | DEC Arm A: 40 mg Cobimetinib + 200 mg Ipatasertib | DEC Arm A: 60 mg Cobimetinib + 200 mg Ipatasertib | DEC Arm A: 60 mg Cobimetinib + 300 mg Ipatasertib | DEC Arm A: 40 mg Cobimetinib + 400 mg Ipatasertib | DEC Arm B: 100 mg Cobimetinib + 200 mg Ipatasertib | DEC Arm B: 125 mg Cobimetinib + 200 mg Ipatasertib | DEC Arm B: 125 mg Cobimetinib + 400 mg Ipatasertib | DEC Arm B: 150 mg Cobimetinib + 300 mg Ipatasertib | DEC Arm B: 175 mg Cobimetinib + 200 mg Ipatasertib | DEC Arm B: 150 mg Cobimetinib + 200 mg Ipatasertib | DEC Arm B: 100 mg Cobimetinib + 400 mg Ipatasertib | Endometrial Carcinoma: 140 mg Cobimetinib + 300 mg Ipatasertib | Breast Cancer: 140 mg Cobimetinib + 300 mg Ipatasertib
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 14 | 5
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 14 | 5
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Not completed — Progression of Disease | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 12 | 4

BASELINE CHARACTERISTICS:
Population: All enrolled participants.
Groups:
- DEC Arm A: 40 mg Cobimetinib + 200 mg Ipatasertib: Participants received oral 40 mg cobimetinib and 200 mg ipatasertib concurrently once daily on Days 1-21, with a 7-day dosing holiday on Days 22-28, every 28 days (1 Cycle=28 Days) until disease progression, unacceptable toxicity, or any other discontinuation criteria were met.
- Total: Total of all reporting groups
Arm/Group | DEC Arm A: 40 mg Cobimetinib + 200 mg Ipatasertib | DEC Arm A: 60 mg Cobimetinib + 200 mg Ipatasertib | DEC Arm A: 60 mg Cobimetinib + 300 mg Ipatasertib | DEC Arm A: 40 mg Cobimetinib + 400 mg Ipatasertib | DEC Arm B: 100 mg Cobimetinib + 200 mg Ipatasertib | DEC Arm B: 125 mg Cobimetinib + 200 mg Ipatasertib | DEC Arm B: 125 mg Cobimetinib + 400 mg Ipatasertib | DEC Arm B: 150 mg Cobimetinib + 300 mg Ipatasertib | DEC Arm B: 175 mg Cobimetinib + 200 mg Ipatasertib | DEC Arm B: 150 mg Cobimetinib + 200 mg Ipatasertib | DEC Arm B: 100 mg Cobimetinib + 400 mg Ipatasertib | Endometrial Carcinoma: 140 mg Cobimetinib + 300 mg Ipatasertib | Breast Cancer: 140 mg Cobimetinib + 300 mg Ipatasertib | Total
Number analyzed (Participants) | 3 | 7 | 3 | 4 | 4 | 4 | 3 | 7 | 3 | 7 | 3 | 14 | 5 | 67
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.0 (3.5) | 59.1 (8.7) | 58.3 (5.5) | 66.8 (16.5) | 62.3 (7.0) | 51.8 (10.9) | 59.0 (9.2) | 58.6 (11.9) | 61.0 (13.7) | 57.6 (10.9) | 52.7 (24.9) | 62.9 (8.7) | 49.0 (10.1) | 59.0 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 1 | 3 | 3 | 4 | 2 | 3 | 2 | 4 | 1 | 14 | 5 | 48
  Male | 1 | 3 | 2 | 1 | 1 | 0 | 1 | 4 | 1 | 3 | 2 | 0 | 0 | 19

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicities (DLTs)
Description: DLT is defined as 1 of the following toxicities considered by the investigator to be possibly related to study drugs: a) Grade (G) ≥3 febrile neutropenia, b) G ≥4 neutropenia (absolute neutrophil count [ANC] <500/ microliter [μL]) lasting >5 days , c) G ≥4 thrombocytopenia lasting >2 days, d) G ≥4 anemia, e) G ≥3 elevation of total bilirubin or hepatic transaminase or alkaline phosphatase (ALP) lasting >3 days, f) Hepatic transaminases >3 × Upper Limit of Normal (ULN) and an increase in total bilirubin >2 × ULN without any findings of cholestasis and in the absence of other contributory factors, g) G ≥2 visual changes that do not resolve to baseline within 14 days, h) 1 episode of fasting G 4 hyperglycemia or 3 episodes of fasting, i) G 3 hyperglycemia on separate days within 7 days, j) G ≥4 fasting hypercholesterolemia or triglyceridemia for ≥2 weeks, k) G ≥3 nausea, vomiting, or diarrhea despite maximal supportive medications lasting for ≥3 days.
Time Frame: Cycle 1 (28 Days)
Population: Safety analysis set included all participants who received at least 1 dose of study treatment. This outcome was analyzed in safety analysis population participants in dose escalation cohorts.
Measure: Number; unit: participants
Arm/Group | DEC Arm A: 40 mg Cobimetinib + 200 mg Ipatasertib | DEC Arm A: 60 mg Cobimetinib + 200 mg Ipatasertib | DEC Arm A: 60 mg Cobimetinib + 300 mg Ipatasertib | DEC Arm A: 40 mg Cobimetinib + 400 mg Ipatasertib | DEC Arm B: 100 mg Cobimetinib + 200 mg Ipatasertib | DEC Arm B: 125 mg Cobimetinib + 200 mg Ipatasertib | DEC Arm B: 125 mg Cobimetinib + 400 mg Ipatasertib | DEC Arm B: 150 mg Cobimetinib + 300 mg Ipatasertib | DEC Arm B: 175 mg Cobimetinib + 200 mg Ipatasertib | DEC Arm B: 150 mg Cobimetinib + 200 mg Ipatasertib | DEC Arm B: 100 mg Cobimetinib + 400 mg Ipatasertib
Number analyzed (Participants) | 3 | 7 | 3 | 4 | 4 | 4 | 3 | 7 | 3 | 6 | 3
participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Number of DLTs Categorized as Per the Nature
Description: DLT is defined as 1 of the following toxicities considered by the investigator to be possibly related to study drugs: a) G ≥3 febrile neutropenia, b) G ≥4 neutropenia (ANC <500/μL) lasting >5 days , c) G ≥4 thrombocytopenia lasting >2 days, d) G ≥4 anemia, e) G ≥3 elevation of total bilirubin or hepatic transaminase or ALP lasting >3 days, f) Hepatic transaminases >3 × ULN and an increase in total bilirubin >2 × ULN without any findings of cholestasis and in the absence of other contributory factors, g) G ≥2 visual changes that do not resolve to baseline within 14 days, h) 1 episode of fasting G 4 hyperglycemia or 3 episodes of fasting, i) G 3 hyperglycemia on separate days within 7 days, j) G ≥4 fasting hypercholesterolemia or triglyceridemia for ≥2 weeks, k) G ≥3 nausea, vomiting, or diarrhea despite maximal supportive medications lasting for ≥3 days. Hematologic, Hepatic and non-hematologic and non-hepatic DLT categories were to be reported.
Time Frame: Cycle 1 (28 Days)
Population: Data for this outcome measure was not analyzed as no participant experienced DLT.
Arm/Group | DEC Arm A: 40 mg Cobimetinib + 200 mg Ipatasertib | DEC Arm A: 60 mg Cobimetinib + 200 mg Ipatasertib | DEC Arm A: 60 mg Cobimetinib + 300 mg Ipatasertib | DEC Arm A: 40 mg Cobimetinib + 400 mg Ipatasertib | DEC Arm B: 100 mg Cobimetinib + 200 mg Ipatasertib | DEC Arm B: 125 mg Cobimetinib + 200 mg Ipatasertib | DEC Arm B: 125 mg Cobimetinib + 400 mg Ipatasertib | DEC Arm B: 150 mg Cobimetinib + 300 mg Ipatasertib | DEC Arm B: 175 mg Cobimetinib + 200 mg Ipatasertib | DEC Arm B: 150 mg Cobimetinib + 200 mg Ipatasertib | DEC Arm B: 100 mg Cobimetinib + 400 mg Ipatasertib
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Maximum Tolerated Doses (MTDs) in Combination of Cobimetinib and Ipatasertib During Dose-Escalation Stage 1
Description: An adverse event (AE) is any unfavorable and unintended sign, symptom, or disease temporally associated with the use of an investigational medicinal product (IMP) or other protocol-imposed intervention, regardless of attribution. On the basis of AEs that did not meet protocol-defined DLT criteria (defined in Outcome measure 1) but indicated intolerability of a given dose combination, the combination MTDs were determined (as per investigator) during Stage 1 of the study.
Time Frame: Cycle 1 (28 Days)
Population: Safety analysis population participants from dose escalation cohorts.
Measure: Number; unit: milligrams
Groups:
- Stage 1 DECs: During Stage 1, participants received cobimetinib and ipatasertib combination doses either under Arm A (21/7 dosing schedule [cobimetinib and ipatasertib taken concurrently once daily on Days 1-21, with a 7-day dosing holiday on Days 22-28, every 28 days]) or under Arm B (intermittent cobimetinib dosing schedule [ipatasertib taken once daily on Days 1-21 consecutively with concurrent dosing of cobimetinib on Days 1, 4, 8, 11, 15, and 18 with a 7-day dosing holiday on Days 22-28, every 28 days)] until disease progression, unacceptable toxicity, or any other discontinuation criteria were met.
Arm/Group | Stage 1 DECs
Number analyzed (Participants) | 48
milligrams
  Arm A Cobimetinib dose | 60
  Arm A Ipatasertib dose | 200
  Arm B Cobimetinib dose | 150
  Arm B Ipatasertib dose | 300

4. Primary Outcome: Number of Participants With At Least One AE Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), Version (V) 4.0
Description: AE was defined in Outcome Measure 3. AEs were graded as per NCI CTCAE V 4.0 as follows: G 1: asymptomatic or mild symptoms, clinical or diagnostic observations only, intervention not indicated; G 2: minimal, local or noninvasive intervention indicated, limiting age-appropriate instrumental activities of daily living (ADL) (instrumental ADL refers to preparing meals, shopping for groceries or clothes, using the telephone, managing money and others); G 3: severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated, disabling, limiting self care ADL (refers to bathing, dressing and undressing, feeding self, using the toilet, taking medications, and not bedridden); G 4: Life-threatening consequences, urgent intervention indicated; G 5: Death related to AE. If a participant had multiple events of different grades, the highest grade that occurred in that participant was counted.
Time Frame: From Baseline up to 30 days after the last dose of study treatment or until initiation of another anticancer treatment whichever occurred first (Up to 33 months)
Population: Safety analysis population.
Measure: Number; unit: participants
Groups:
- DECs and Expansion Cohorts: Included all participants who were treated under Stage 1 (Dose Escalation Cohorts) and Stage 2 (Dose Expansion Cohorts).
Arm/Group | DECs and Expansion Cohorts
Number analyzed (Participants) | 66
participants
  Grade 1 (G 1) | 4
  Grade 2 (G 2) | 15
  Grade 3 (G 3) | 36
  Grade 4 (G 4) | 1
  Grade 5 (G 5) | 10

5. Secondary Outcome: Area Under Concentration-Time Curve From Time Zero to Last Measurable Concentration After Dose [AUC0-Last] of Ipatasertib and Cobimetinib on Day 1 and Day 15
Time Frame: Predose (0 hour), 1, 2, 4, 6 and 24 hours postdose on Day 1 and Day 15 of Cycle 1
Population: Pharmacokinetic analysis population: Included all participants who received study treatment and had at least 1 cobimetinib and ipatasertib plasma concentration available. "n" represents the number of participants who were evaluable for that particular assessment.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hours/milliliter (ng*h/mL)
Arm/Group | DEC Arm A: 40 mg Cobimetinib + 200 mg Ipatasertib | DEC Arm A: 60 mg Cobimetinib + 200 mg Ipatasertib | DEC Arm A: 60 mg Cobimetinib + 300 mg Ipatasertib | DEC Arm A: 40 mg Cobimetinib + 400 mg Ipatasertib | DEC Arm B: 100 mg Cobimetinib + 200 mg Ipatasertib | DEC Arm B: 125 mg Cobimetinib + 200 mg Ipatasertib | DEC Arm B: 125 mg Cobimetinib + 400 mg Ipatasertib | DEC Arm B: 150 mg Cobimetinib + 300 mg Ipatasertib | DEC Arm B: 175 mg Cobimetinib + 200 mg Ipatasertib | DEC Arm B: 150 mg Cobimetinib + 200 mg Ipatasertib | DEC Arm B: 100 mg Cobimetinib + 400 mg Ipatasertib | Endometrial Carcinoma: 140 mg Cobimetinib + 300 mg Ipatasertib | Breast Cancer: 140 mg Cobimetinib + 300 mg Ipatasertib
Number analyzed (Participants) | 3 | 7 | 2 | 4 | 4 | 4 | 3 | 6 | 2 | 6 | 2 | 14 | 5
nanograms*hours/milliliter (ng*h/mL)
  Ipatasertib Day 1 (n=3,7,1,4,4,4,3,5,2,6,2,14,5) | 688 (106) | 538 (33.8) | 1760 (NA) — As n=1, geometric coefficient of variation is not applicable | 2170 (74.9) | 255 (203) | 956 (43.5) | 1420 (46.4) | 790 (78.8) | 838 (239) | 424 (67.9) | 2030 (46.4) | 1450 (48.7) | 1540 (11.3)
  Ipatasertib Day 15 (n=3,6,2,1,4,3,1,6,2,5,2,7,2) | 703 (40.8) | 781 (20.7) | 2440 (45.2) | 1750 (NA) — As n=1, geometric coefficient of variation is not applicable | 599 (133) | 1760 (62.3) | 2230 (NA) — As n=1, geometric coefficient of variation is not applicable | 1260 (85.2) | 668 (148) | 866 (58.1) | 3390 (9.70) | 1070 (65.2) | 1270 (13.3)
  Cobimetinib Day 1 (n=3,7,1,4,4,4,3,5,2,6,2,14,5) | 1500 (320) | 1130 (68.6) | 5050 (NA) — As n=1, geometric coefficient of variation is not applicable | 1920 (87.8) | 3740 (139) | 5580 (54.4) | 2690 (50.7) | 2710 (60.7) | 13600 (111) | 3270 (89.2) | 4330 (39.3) | 11400 (64.1) | 10800 (41.0)
  Cobimetinib Day 15 (n=3,6,2,1,4,3,1,6,1,5,2,7,2) | 3250 (223) | 3260 (48.6) | 7080 (91.1) | 2500 (NA) — As n=1, geometric coefficient of variation is not applicable | 3230 (96.8) | 8140 (5.65) | 4400 (NA) — As n=1, geometric coefficient of variation is not applicable | 4970 (65.5) | 8570 (NA) — As n=1, geometric coefficient of variation is not applicable | 3980 (111) | 6830 (38.4) | 8880 (64.8) | 1480 (10800)

6. Secondary Outcome: Maximum Plasma Concentration (Cmax) of Ipatasertib and Cobimetinib on Day 1 and Day 15
Time Frame: Predose (0 hour), 1, 2, 4, 6 and 24 hours postdose on Day 1 and Day 15 of Cycle 1
Population: Pharmacokinetic analysis population. "n" represents the number of participants who were evaluable for that particular assessment.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Arm/Group | DEC Arm A: 40 mg Cobimetinib + 200 mg Ipatasertib | DEC Arm A: 60 mg Cobimetinib + 200 mg Ipatasertib | DEC Arm A: 60 mg Cobimetinib + 300 mg Ipatasertib | DEC Arm A: 40 mg Cobimetinib + 400 mg Ipatasertib | DEC Arm B: 100 mg Cobimetinib + 200 mg Ipatasertib | DEC Arm B: 125 mg Cobimetinib + 200 mg Ipatasertib | DEC Arm B: 125 mg Cobimetinib + 400 mg Ipatasertib | DEC Arm B: 150 mg Cobimetinib + 300 mg Ipatasertib | DEC Arm B: 175 mg Cobimetinib + 200 mg Ipatasertib | DEC Arm B: 150 mg Cobimetinib + 200 mg Ipatasertib | DEC Arm B: 100 mg Cobimetinib + 400 mg Ipatasertib | Endometrial Carcinoma: 140 mg Cobimetinib + 300 mg Ipatasertib | Breast Cancer: 140 mg Cobimetinib + 300 mg Ipatasertib
Number analyzed (Participants) | 3 | 7 | 2 | 4 | 4 | 4 | 3 | 6 | 2 | 6 | 2 | 14 | 5
nanograms per milliliter (ng/mL)
  Ipatasertib Day 1 (n=3,7,1,4,4,4,3,5,2,6,2,14,5) | 137 (244) | 97.1 (92.2) | 300 (NA) — As n=1, geometric coefficient of variation is not applicable | 336 (118) | 42.9 (560) | 156 (32.8) | 329 (104) | 141 (34.3) | 99.9 (254) | 95.8 (57.1) | 262 (122) | 268 (48.3) | 374 (48.2)
  Ipatasertib Day 15 (n=3,6,2,1,4,3,1,6,2,5,2,7,2) | 94.5 (55.0) | 130 (47.1) | 386 (58.4) | 137 (NA) — As n=1, geometric coefficient of variation is not applicable | 86.9 (237) | 165 (33.9) | 441 (NA) — As n=1, geometric coefficient of variation is not applicable | 170 (64.4) | 72.9 (200) | 114 (53.9) | 450 (16.9) | 149 (113) | 156 (12.7)
  Cobimetinib Day 1 (n=3,7,1,4,4,4,3,5,2,6,2,14,5) | 134 (333) | 78.6 (73.2) | 312 (NA) — As n=1, geometric coefficient of variation is not applicable | 109 (85.4) | 259 (192) | 405 (45.9) | 192 (50.3) | 220 (64.9) | 1040 (151) | 262 (59.9) | 249 (46.0) | 799 (55.8) | 840 (56.6)
  Cobimetinib Day 15 (n=3,6,2,1,4,3,1,6,1,5,2,7,2) | 222 (182) | 215 (61.4) | 407 (72.6) | 121 (NA) — As n=1, geometric coefficient of variation is not applicable | 217 (135) | 511 (14.6) | 376 (NA) — As n=1, geometric coefficient of variation is not applicable | 320 (64.5) | 481 (NA) — As n=1, geometric coefficient of variation is not applicable | 253 (103) | 420 (41.4) | 704 (75.2) | 84.2 (7940)

7. Secondary Outcome: Time Taken to Reach Cmax (Tmax) of Ipatasertib and Cobimetinib on Day 1 and Day 15
Time Frame: Predose (0 hour), 1, 2, 4, 6 and 24 hours postdose on Day 1 and Day 15 of Cycle 1
Population: as for outcome 6
Measure: Median (Full Range); unit: hours
Arm/Group | DEC Arm A: 40 mg Cobimetinib + 200 mg Ipatasertib | DEC Arm A: 60 mg Cobimetinib + 200 mg Ipatasertib | DEC Arm A: 60 mg Cobimetinib + 300 mg Ipatasertib | DEC Arm A: 40 mg Cobimetinib + 400 mg Ipatasertib | DEC Arm B: 100 mg Cobimetinib + 200 mg Ipatasertib | DEC Arm B: 125 mg Cobimetinib + 200 mg Ipatasertib | DEC Arm B: 125 mg Cobimetinib + 400 mg Ipatasertib | DEC Arm B: 150 mg Cobimetinib + 300 mg Ipatasertib | DEC Arm B: 175 mg Cobimetinib + 200 mg Ipatasertib | DEC Arm B: 150 mg Cobimetinib + 200 mg Ipatasertib | DEC Arm B: 100 mg Cobimetinib + 400 mg Ipatasertib | Endometrial Carcinoma: 140 mg Cobimetinib + 300 mg Ipatasertib | Breast Cancer: 140 mg Cobimetinib + 300 mg Ipatasertib
Number analyzed (Participants) | 3 | 7 | 2 | 4 | 4 | 4 | 3 | 6 | 2 | 6 | 2 | 14 | 5
hours
  Ipatasertib Day 1 (n=3,7,1,4,4,4,3,5,2,6,2,14,5) | 1.03 [1.00 to 1.05] | 1.02 [0.92 to 4.08] | 1.00 [NA to NA] — As n=1, full range is not applicable | 1.04 [1.00 to 4.08] | 1.00 [0.92 to 4.78] | 3.04 [1.00 to 4.13] | 1.00 [0.90 to 2.40] | 2.00 [1.92 to 4.00] | 3.17 [2.08 to 4.25] | 1.08 [1.00 to 2.00] | 1.52 [1.00 to 2.03] | 1.47 [0.95 to 4.00] | 1.00 [1.00 to 1.00]
  Ipatasertib Day 15 (n=3,6,2,1,4,3,1,6,2,5,2,7,2) | 2.03 [0.95 to 2.25] | 1.03 [1.00 to 3.83] | 1.04 [1.00 to 1.08] | 6.05 [NA to NA] — As n=1, full range is not applicable | 1.04 [1.00 to 1.15] | 1.00 [1.00 to 2.00] | 1.00 [NA to NA] — As n=1, full range is not applicable | 1.19 [1.00 to 6.00] | 1.57 [1.00 to 2.13] | 1.00 [0.92 to 4.08] | 0.98 [0.93 to 1.02] | 1.08 [0.92 to 3.58] | 0.97 [0.93 to 1.00]
  Cobimetinib Day 1 (n=3,7,1,4,4,4,3,5,2,6,2,14,5) | 2.00 [2.00 to 4.00] | 3.97 [1.92 to 24.0] | 2.05 [NA to NA] — As n=1, full range is not applicable | 3.83 [2.02 to 5.95] | 3.04 [2.00 to 6.00] | 3.03 [2.00 to 6.00] | 4.05 [4.00 to 4.27] | 4.00 [2.00 to 23.9] | 24.0 [22.0 to 26.0] | 3.91 [2.00 to 4.25] | 5.92 [5.83 to 6.00] | 3.08 [1.00 to 24.4] | 2.08 [2.00 to 5.42]
  Cobimetinib Day 15 (n=3,6,2,1,4,3,1,6,1,5,2,7,2) | 2.25 [2.00 to 4.00] | 3.92 [2.08 to 4.00] | 3.01 [2.00 to 4.02] | 6.05 [NA to NA] — As n=1, full range is not applicable | 4.78 [1.15 to 5.97] | 4.03 [4.00 to 24.2] | 1.88 [NA to NA] — As n=1, full range is not applicable | 4.06 [2.25 to 23.7] | 5.92 [NA to NA] — As n=1, full range is not applicable | 4.00 [0.00 to 5.58] | 13.1 [2.00 to 24.1] | 2.00 [1.00 to 24.3] | 1.96 [1.92 to 2.00]

8. Secondary Outcome: Last Measurable Concentration (Clast) of Ipatasertib and Cobimetinib on Day 1 and Day 15
Time Frame: Predose (0 hour), 1, 2, 4, 6 and 24 hours postdose on Day 1 and Day 15 of Cycle 1
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | DEC Arm A: 40 mg Cobimetinib + 200 mg Ipatasertib | DEC Arm A: 60 mg Cobimetinib + 200 mg Ipatasertib | DEC Arm A: 60 mg Cobimetinib + 300 mg Ipatasertib | DEC Arm A: 40 mg Cobimetinib + 400 mg Ipatasertib | DEC Arm B: 100 mg Cobimetinib + 200 mg Ipatasertib | DEC Arm B: 125 mg Cobimetinib + 200 mg Ipatasertib | DEC Arm B: 125 mg Cobimetinib + 400 mg Ipatasertib | DEC Arm B: 150 mg Cobimetinib + 300 mg Ipatasertib | DEC Arm B: 175 mg Cobimetinib + 200 mg Ipatasertib | DEC Arm B: 150 mg Cobimetinib + 200 mg Ipatasertib | DEC Arm B: 100 mg Cobimetinib + 400 mg Ipatasertib | Endometrial Carcinoma: 140 mg Cobimetinib + 300 mg Ipatasertib | Breast Cancer: 140 mg Cobimetinib + 300 mg Ipatasertib
Number analyzed (Participants) | 3 | 7 | 2 | 4 | 4 | 4 | 3 | 6 | 2 | 6 | 2 | 14 | 5
ng/mL
  Ipatasertib Day 1 (n=3,7,1,4,4,4,3,5,2,6,2,14,5) | 6.18 (4.90) | 6.07 (1.99) | 23.7 (NA) — As n=1, standard deviation is not applicable | 25.1 (11.3) | 4.32 (2.60) | 13.4 (8.29) | 15.2 (5.15) | 7.05 (11.60) | 18.2 (16.2) | 6.00 (4.18) | 30.0 (5.66) | 18.0 (10.1) | 15.4 (6.38)
  Ipatasertib Day 15 (n=3,6,2,1,4,3,1,6,2,5,2,7,2) | 14.1 (4.54) | 11.6 (1.79) | 38.0 (14.5) | 30.6 (NA) — As n=1, standard deviation is not applicable | 12.8 (6.85) | 30.6 (22.2) | 39.3 (NA) — As n=1, standard deviation is not applicable | 21.90 (45.50) | 13.0 (7.66) | 16.9 (10.9) | 54.7 (15.5) | 20.7 (12.1) | 14.5 (8.68)
  Cobimetinib Day 1 (n=3,7,1,4,4,4,3,5,2,6,2,14,5) | 79.4 (119) | 35.9 (10.5) | 150 (NA) — As n=1, standard deviation is not applicable | 71.9 (44.0) | 122 (76.5) | 204 (172) | 72.6 (30.7) | 145 (159) | 1280 (1120) | 125 (127) | 160 (17.7) | 386 (237) | 268 (146)
  Cobimetinib Day 15 (n=3,6,2,1,4,3,1,6,1,5,2,7,2) | 228 (319) | 105 (58.3) | 251 (192) | 93.8 (NA) — As n=1, standard deviation is not applicable | 123 (70.2) | 294 (158) | 127 (NA) — As n=1, standard deviation is not applicable | 186 (116) | 283 (NA) — As n=1, standard deviation is not applicable | 204 (254) | 280 (53.0) | 299 (172) | 227 (316)

9. Secondary Outcome: Number of Participants With Objective Response of Complete Response (CR) or Partial Response (PR) According to Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1)
Description: RECIST v1.1 (for measurable disease), CR: disappearance of all target lesions, reduction in short axis <10 millimeters in pathological lymph nodes (target and non-target lesions); PR: at least a 30 percent (%) decrease in the sum of the longest diameter of target lesions, taking as reference the baseline sum longest diameter. Responses were confirmed by repeat assessments ≥4 weeks after initial documentation.
Time Frame: Screening, Days 21-28 of Cycle 2, Day 25 (± 3 days) of Cycle 4 and every 8 weeks thereafter till study completion (Up to 33 months)
Population: Safety analysis population.
Measure: Number; unit: participants
Arm/Group | DEC Arm A: 40 mg Cobimetinib + 200 mg Ipatasertib | DEC Arm A: 60 mg Cobimetinib + 200 mg Ipatasertib | DEC Arm A: 60 mg Cobimetinib + 300 mg Ipatasertib | DEC Arm A: 40 mg Cobimetinib + 400 mg Ipatasertib | DEC Arm B: 100 mg Cobimetinib + 200 mg Ipatasertib | DEC Arm B: 125 mg Cobimetinib + 200 mg Ipatasertib | DEC Arm B: 125 mg Cobimetinib + 400 mg Ipatasertib | DEC Arm B: 150 mg Cobimetinib + 300 mg Ipatasertib | DEC Arm B: 175 mg Cobimetinib + 200 mg Ipatasertib | DEC Arm B: 150 mg Cobimetinib + 200 mg Ipatasertib | DEC Arm B: 100 mg Cobimetinib + 400 mg Ipatasertib | Endometrial Carcinoma: 140 mg Cobimetinib + 300 mg Ipatasertib | Breast Cancer: 140 mg Cobimetinib + 300 mg Ipatasertib
Number analyzed (Participants) | 3 | 7 | 3 | 4 | 4 | 4 | 3 | 7 | 3 | 6 | 3 | 14 | 5
participants | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0

10. Secondary Outcome: Duration of Objective Response for Participants With Measurable Disease According to RECIST v1.1
Description: Duration of response, defined as the time from first occurrence of a documented objective response until the time of disease progression, as determined by investigator review of tumor assessments using RECIST 1.1, or death from any cause during the study (i.e., within 30 days after the last dose of study treatment).
Time Frame: as for outcome 9
Population: This outcome measure was not analyzed as per changes in planned analysis due to very few participants with measurable response.
Arm/Group | DEC Arm A: 40 mg Cobimetinib + 200 mg Ipatasertib | DEC Arm A: 60 mg Cobimetinib + 200 mg Ipatasertib | DEC Arm A: 60 mg Cobimetinib + 300 mg Ipatasertib | DEC Arm A: 40 mg Cobimetinib + 400 mg Ipatasertib | DEC Arm B: 100 mg Cobimetinib + 200 mg Ipatasertib | DEC Arm B: 125 mg Cobimetinib + 200 mg Ipatasertib | DEC Arm B: 125 mg Cobimetinib + 400 mg Ipatasertib | DEC Arm B: 150 mg Cobimetinib + 300 mg Ipatasertib | DEC Arm B: 175 mg Cobimetinib + 200 mg Ipatasertib | DEC Arm B: 150 mg Cobimetinib + 200 mg Ipatasertib | DEC Arm B: 100 mg Cobimetinib + 400 mg Ipatasertib | Endometrial Carcinoma: 140 mg Cobimetinib + 300 mg Ipatasertib | Breast Cancer: 140 mg Cobimetinib + 300 mg Ipatasertib
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

11. Secondary Outcome: Progression-Free Survival (PFS) Time for Participants With Measurable Disease According to RECIST v1.1
Description: PFS is defined as the time from study treatment initiation to the first occurrence of disease progression, as determined by investigator review of tumor assessments using RECIST 1.1, or death from any cause during the study (i.e., within 30 days after the last dose of study treatment).
Time Frame: as for outcome 9
Population: as for outcome 10
Arm/Group | DEC Arm A: 40 mg Cobimetinib + 200 mg Ipatasertib | DEC Arm A: 60 mg Cobimetinib + 200 mg Ipatasertib | DEC Arm A: 60 mg Cobimetinib + 300 mg Ipatasertib | DEC Arm A: 40 mg Cobimetinib + 400 mg Ipatasertib | DEC Arm B: 100 mg Cobimetinib + 200 mg Ipatasertib | DEC Arm B: 125 mg Cobimetinib + 200 mg Ipatasertib | DEC Arm B: 125 mg Cobimetinib + 400 mg Ipatasertib | DEC Arm B: 150 mg Cobimetinib + 300 mg Ipatasertib | DEC Arm B: 175 mg Cobimetinib + 200 mg Ipatasertib | DEC Arm B: 150 mg Cobimetinib + 200 mg Ipatasertib | DEC Arm B: 100 mg Cobimetinib + 400 mg Ipatasertib | Endometrial Carcinoma: 140 mg Cobimetinib + 300 mg Ipatasertib | Breast Cancer: 140 mg Cobimetinib + 300 mg Ipatasertib
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From Baseline up to 30 days after the last dose of study treatment or until initiation of another anticancer treatment whichever occurred first (Up to 33 months)
Arm/Group | DEC Arm A: 40 mg Cobimetinib + 200 mg Ipatasertib | DEC Arm A: 60 mg Cobimetinib + 200 mg Ipatasertib | DEC Arm A: 60 mg Cobimetinib + 300 mg Ipatasertib | DEC Arm A: 40 mg Cobimetinib + 400 mg Ipatasertib | DEC Arm B: 100 mg Cobimetinib + 200 mg Ipatasertib | DEC Arm B: 125 mg Cobimetinib + 200 mg Ipatasertib | DEC Arm B: 125 mg Cobimetinib + 400 mg Ipatasertib | DEC Arm B: 150 mg Cobimetinib + 300 mg Ipatasertib | DEC Arm B: 175 mg Cobimetinib + 200 mg Ipatasertib | DEC Arm B: 150 mg Cobimetinib + 200 mg Ipatasertib | DEC Arm B: 100 mg Cobimetinib + 400 mg Ipatasertib | Endometrial Carcinoma: 140 mg Cobimetinib + 300 mg Ipatasertib | Breast Cancer: 140 mg Cobimetinib + 300 mg Ipatasertib
Serious Adverse Events (participants affected / at risk) | 1/3 | 2/7 | 0/3 | 2/4 | 1/4 | 3/4 | 1/3 | 1/7 | 0/3 | 2/6 | 2/3 | 10/14 | 2/5
Other Adverse Events (participants affected / at risk) | 3/3 | 7/7 | 3/3 | 4/4 | 4/4 | 4/4 | 3/3 | 7/7 | 3/3 | 6/6 | 3/3 | 14/14 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DEC Arm A: 40 mg Cobimetinib + 200 mg Ipatasertib (N=3) | DEC Arm A: 60 mg Cobimetinib + 200 mg Ipatasertib (N=7) | DEC Arm A: 60 mg Cobimetinib + 300 mg Ipatasertib (N=3) | DEC Arm A: 40 mg Cobimetinib + 400 mg Ipatasertib (N=4) | DEC Arm B: 100 mg Cobimetinib + 200 mg Ipatasertib (N=4) | DEC Arm B: 125 mg Cobimetinib + 200 mg Ipatasertib (N=4) | DEC Arm B: 125 mg Cobimetinib + 400 mg Ipatasertib (N=3) | DEC Arm B: 150 mg Cobimetinib + 300 mg Ipatasertib (N=7) | DEC Arm B: 175 mg Cobimetinib + 200 mg Ipatasertib (N=3) | DEC Arm B: 150 mg Cobimetinib + 200 mg Ipatasertib (N=6) | DEC Arm B: 100 mg Cobimetinib + 400 mg Ipatasertib (N=3) | Endometrial Carcinoma: 140 mg Cobimetinib + 300 mg Ipatasertib (N=14) | Breast Cancer: 140 mg Cobimetinib + 300 mg Ipatasertib (N=5)
Atrial Fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Intestinal Obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Large Intestinal Obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Small Intestinal Obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Disease Progression (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bile Duct Obstruction (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Clostridium Difficile Colitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hip Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Toxicity to Various Agents (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Liver Function Test Abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Malignant Neoplasm Progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mental Status Changes (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Renal Failure (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Renal Failure Acute (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DEC Arm A: 40 mg Cobimetinib + 200 mg Ipatasertib (N=3) | DEC Arm A: 60 mg Cobimetinib + 200 mg Ipatasertib (N=7) | DEC Arm A: 60 mg Cobimetinib + 300 mg Ipatasertib (N=3) | DEC Arm A: 40 mg Cobimetinib + 400 mg Ipatasertib (N=4) | DEC Arm B: 100 mg Cobimetinib + 200 mg Ipatasertib (N=4) | DEC Arm B: 125 mg Cobimetinib + 200 mg Ipatasertib (N=4) | DEC Arm B: 125 mg Cobimetinib + 400 mg Ipatasertib (N=3) | DEC Arm B: 150 mg Cobimetinib + 300 mg Ipatasertib (N=7) | DEC Arm B: 175 mg Cobimetinib + 200 mg Ipatasertib (N=3) | DEC Arm B: 150 mg Cobimetinib + 200 mg Ipatasertib (N=6) | DEC Arm B: 100 mg Cobimetinib + 400 mg Ipatasertib (N=3) | Endometrial Carcinoma: 140 mg Cobimetinib + 300 mg Ipatasertib (N=14) | Breast Cancer: 140 mg Cobimetinib + 300 mg Ipatasertib (N=5)
Anaemia (Blood and lymphatic system disorders) | 1 | 4 | 1 | 1 | 3 | 3 | 0 | 0 | 1 | 1 | 2 | 6 | 1
Anaemia Vitamin B12 Deficiency (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypercoagulation (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 3 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 2 | 0
Atrial Fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atrial Flutter (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Palpitations (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinus Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinus Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Supraventricular Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Eye Discharge (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye Disorder (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Eye Pain (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lacrimation Increased (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ocular Hyperaemia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Periorbital Oedema (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Photopsia (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vision Blurred (Eye disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 0 | 1 | 1
Visual Acuity Reduced Transiently (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Visual Impairment (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Vitreous Floaters (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Abdominal Discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0
Abdominal Distension (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 3 | 0
Abdominal Pain (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 0 | 1 | 1 | 2 | 0 | 2 | 1 | 3 | 1
Abdominal Pain Lower (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Anal Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Aphthous Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Ascites (Gastrointestinal disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Chapped Lips (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 4 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 5 | 2
Diarrhoea (Gastrointestinal disorders) | 3 | 6 | 3 | 4 | 4 | 3 | 3 | 7 | 3 | 4 | 3 | 14 | 5
Dry Mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 1 | 0 | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1
Eructation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 0
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ileus Paralytic (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lip Dry (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lip Oedema (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 4 | 2 | 4 | 3 | 2 | 1 | 4 | 1 | 6 | 3 | 11 | 4
Obstruction Gastric (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Oesophageal Pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral Pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oral Pruritus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Paraesthesia Oral (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Peptic Ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Retching (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 5 | 1
Tongue Oedema (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 4 | 2 | 4 | 3 | 3 | 2 | 3 | 2 | 5 | 3 | 12 | 3
Asthenia (General disorders) | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 4 | 4
Catheter Site Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Chest Pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Chills (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Early Satiety (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Face Oedema (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Fatigue (General disorders) | 3 | 3 | 1 | 2 | 2 | 1 | 2 | 4 | 1 | 4 | 3 | 5 | 1
Gait Disturbance (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Medical Device Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Mucosal inflammation (General disorders) | 0 | 3 | 0 | 2 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 1 | 0
Non-cardiac Chest Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Oedema Peripheral (General disorders) | 2 | 2 | 0 | 2 | 3 | 2 | 0 | 2 | 0 | 1 | 0 | 1 | 1
Pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Peripheral Swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 1 | 1 | 1 | 1 | 0 | 1 | 0 | 1 | 1 | 1 | 0
Systemic Inflammatory Response Syndrome (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Contrast Media Allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Acute Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Candida Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Clostridium Difficile Colitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hordeolum (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infected Skin Ulcer (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Localised Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Mucosal Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Oral Candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Paronychia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Urinary Tract Infection (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 0 | 1 | 1 | 1 | 3 | 1
Vaginal Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Viral Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Animal Bite (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Alanine Aminotransferase Increased (Investigations) | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 1 | 1
Amylase Increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Aspartate Aminotransferase Increased (Investigations) | 0 | 2 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 1 | 1 | 2 | 1
Blood Alkaline Phosphatase (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood Alkaline Phosphatase Increased (Investigations) | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0
Blood Calcium Decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood Chloride Decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood Cholesterol Increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood Creatine Phosphokinase Increased (Investigations) | 2 | 3 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 1 | 0
Blood Creatinine Decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood Creatinine Increased (Investigations) | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 2 | 1 | 0
Blood Glucose Increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood Insulin Increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0
Blood Lactate Dehydrogenase Increased (Investigations) | 1 | 2 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 0
Blood Sodium Decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood Urea Decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood Urea Increased (Investigations) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Blood Uric Acid Increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Carbohydrate Antigen 15-3 Increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Carbon Dioxide Decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac Murmur (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Electrocardiogram QT Prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Heart Rate Increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
High Density Lipoprotein Decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Insulin C-peptide Increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0
Lipase Increased (Investigations) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lymphocyte Count Decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Monocyte Count Increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neutrophil Count Increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oxygen Saturation Decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Protein Total Increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urine Output Decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Weight Decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
White Blood Cell Count Decreased (Investigations) | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
White Blood Cell Count Increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 1 | 4 | 0 | 1 | 2 | 2 | 0 | 0 | 1 | 1 | 3 | 7 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 1 | 1 | 1 | 1 | 2 | 1 | 0 | 1 | 1 | 1 | 4 | 1
Gout (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 2 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 1 | 1 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 2 | 0 | 1 | 0 | 1 | 1 | 1 | 5 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 5 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 1 | 0 | 0 | 3 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 2 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Salt Craving (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 2 | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 0
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Flank Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Groin Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 1 | 0 | 0 | 0 | 2 | 2
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Depressed Level of Consciousness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Disturbance in Attention (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 1 | 1 | 1 | 0 | 1 | 2
Dysgeusia (Nervous system disorders) | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 2 | 2 | 1 | 2
Headache (Nervous system disorders) | 0 | 2 | 1 | 0 | 2 | 1 | 1 | 1 | 0 | 1 | 0 | 2 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Memory Impairment (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Migraine with Aura (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Monoplegia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Polyneuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Visual Field Defect (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Confusional State (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hallucination (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hallucination, Visual (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 2 | 0
Mental Status Changes (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bladder Spasm (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chromaturia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Incontinence (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Micturition Urgency (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oliguria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0
Renal Failure (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Renal Failure Acute (Renal and urinary disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oedema Genital (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pelvic Pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus Genital (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vaginal Discharge (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vaginal Haemorrhage (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 1 | 2 | 2 | 1 | 1 | 0 | 1 | 0 | 1 | 2
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0
Nasal Discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Painful Respiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Throat Irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Upper-airway Cough Syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Decubitus Ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis Acneiform (Skin and subcutaneous tissue disorders) | 0 | 2 | 2 | 1 | 1 | 2 | 1 | 7 | 3 | 5 | 1 | 8 | 2
Dry Skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nail Discolouration (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 3 | 1
Rash Erythematous (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash Generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Rash Macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash Maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 0 | 1 | 1 | 3 | 0 | 3 | 2 | 2 | 0
Rash Pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin Disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sinus Operation (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Deep Vein Thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Embolism (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Flushing (Vascular disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Hot Flush (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Lymphoedema (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Subclavian Vein Thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0

LIMITATIONS AND CAVEATS:
As per changes in the planned analysis, PFS and duration of response outcome measures were not analyzed as only few participants experienced a measurable response.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.